CLINICAL TRIAL: NCT04895566
Title: Phase 0/1 Topical Application of the Monoclonal Antibody (Mab) sB24M in Patients With Severe Pyoderma
Brief Title: Phase 0/1 Local Application of the Monoclonal Antibody (Mab) sB24M in Patients With Purulent Pyoderma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: SWISS BIOPHARMA MED GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBPM0311m
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Pyoderma; Pyoderma Gangrenosum; Pyoderma Vegetans; Pyoderma Gangrenosum Surrounding Surgical Stoma
MeSH Terms: conditions — Pyoderma; Pyoderma Gangrenosum | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Masking Description: This trial is an open-label, Phase 0, a non-randomized trial that will enroll up to 10 participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- monoclonal antibody (Mab) sB24M (Experimental): Therapy by injecting 200 mg of the monoclonal antibody (Mab) sB24M into the areas affected by pyoderma
  Interventions: Biological: Monoclonal antibody (Mab) sB24M

INTERVENTIONS:
Biological: Monoclonal antibody (Mab) sB24M — 200 mg monoclonal antibody (Mab) sB24 by injection into the affected areas.
  Other Names: CD47 / TNF-α Monoclonal antibody

SUMMARY:
Phase 0/1 local application of the monoclonal antibody (Mab) sB24M in patients with purulent pyoderma (chronic ulcerative pyoderma) by injection into the affected areas.

Monoclonal antibody (Mab) sB24 negatively regulates immune-inflammatory processes through CD47 / TNF-α Axis promotes epithelialization of damaged tissue.

DETAILED DESCRIPTION:
This is an open-label Phase 0 trial that will enroll up to 10 participants with purulent pyoderma (chronic ulcerative pyoderma) by injecting 200 mg of the monoclonal antibody (Mab) sB24M into the areas affected by pyoderma.

Monoclonal antibody (Mab) sB24 negatively regulates immune-inflammatory processes through CD47 / TNF-α Axis promotes epithelialization of damaged tissue.

This study is a first-in-man since previously no Clinical Studies on the local application (injections) of monoclonal antibodies in pyoderma gangrenosum have been conducted.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed severe form of any type of pyoderma with lesions of the skin and muscle tissue was diagnosed
* Male or female, age ≥ 21 years
* Previous treatment with TNF antagonists (infliximab, adalimumab, etanercept, certolizumab, golimumab) ended no earlier than 30 days before starting therapy
* Secondary treatment failure with up to one previous TNFα antagonist treatment (from the list above)
* Secondary failure of corticosteroid treatment
* Adequate hematologic, hepatic, and renal function
* Written informed consent.

Exclusion Criteria:

* History of primary resistance or intolerance to any TNFα antagonist.
* History of congestive heart failure or current, controlled or uncontrolled
* Women who are pregnant or breastfeeding, or women of childbearing age if no effective method of contraception has been used during and for 3 months after the trial
* Men, if no effective contraceptive method was used during the study and for 3 months afterward
* Any prior exposure to Hu5F9-G4 or other CD47 targeting agents
* Previous allogeneic stem cell transplant within 6 months prior to enrollment, active graft versus host disease (GVHD), or need for graft-associated immunosuppression
* Refusal to sign the informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) in patients with severe pyoderma | Approximately 1 year
  The ORR is defined as the percentage of participants who had a confirmed Complete Response or Partial Response using RECIST 1.1

SECONDARY OUTCOMES:
Duration of response (DoR) of patients with severe forms of pyoderma | Approximately 1 year
  The DoR is defined as the time from the first registration of the onset of visible epithelialization of damaged tissues to the first recorded progression of pyoderma

OTHER OUTCOMES:
Evaluation of genetic factors for severe forms of pyoderma. | Approximately 1 year
  Comparative analysis of gene expression in severe forms of pyoderma by partial genome sequencing prior to treatment
Effect of sB24M monoclonal antibody (Mab) therapy on the expression of certain genes in severe forms of pyoderma | Approximately 1 year
  Comparative analysis of gene expression in severe forms of pyoderma by partial genome sequencing before treatment and after three courses of local injections of monoclonal antibody (Mab) sB24M into the areas affected by pyoderma

CONTACTS AND LOCATIONS:
Locations (2):
- Contract Research Organization, Minsk, Belarus
- Contract Research Organization, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: within three months after the end of the trial
URL: https://sbpm.swiss/